CLINICAL TRIAL: NCT03657576
Title: A Phase I Trial of IRS-1 HSV C134 Administered Intratumorally in Patients With Recurrent Malignant Glioma
Brief Title: Trial of C134 in Patients With Recurrent GBM
Acronym: C134-HSV-1
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Gateway for Cancer Research (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, James Markert, MD, Principal Investigator, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: IRB-3000000571; R01CA222903 (NIH)
Record Dates: First submitted 2018-08-21; First posted 2018-09-05 (Actual); Results first posted 2025-07-03 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Glioblastoma Multiforme of Brain; Anaplastic Astrocytoma of Brain; Gliosarcoma of Brain
Keywords: oncolytic virus; glioma; glioblastoma; GBM; HSV; immunotherapy; Brain Tumors
MeSH Terms: conditions — Glioma; Glioblastoma; Brain Neoplasms

STUDY DESIGN:
Intervention Model Description: Modified continuous reassessment model (mCRM). Using this statistical method, dose changes occur based upon toxicities (or lack thereof) observed after a 24 day observation period for the initial dose level. If toxicities occurring at any dose were acceptable, doses for subsequent cohorts can be increased by up to 1 log until a maximum tolerated dose is reached. If toxicities are unacceptable then dose de-escalation occurs until a safe acceptable maximum tolerated dosage is defined. However, it should be noted that the dose alterations are not predictable and cannot be predefined, they are statistically determined after each patient using mCRM software.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- C134 Treatment (Experimental): All patients who enroll will receive C134 inoculation into their tumor (one time procedure with 1-5 inoculation sites)
  Interventions: Biological: C134

INTERVENTIONS:
Biological: C134 — C134 is a virus that was created from an oncolytic Herpes Simplex Virus (oHSV) known to infect and kill tumor cells. The Investigators have made changes to the original virus to make C134. It efficiently infects tumor cells (not normal healthy cells) and induces an immune response to fight the cancer as well.

SUMMARY:
The purpose of this project is to obtain safety information in small groups of individuals, scheduled to receive escalating doses of C134, a cancer killing virus (HSV-1) that has been genetically engineered to safely replicate and kill glioma tumor cells. Safety will be assessed at each dose level before proceeding to the next dose level. A special statistical technique called the Continual Reassessment Method (CRM) will be used to determine when higher doses of virus can be administered. Other objectives of the study include characterization of the activity of C134 after inoculation into the tumor and of the local and systemic immune responses to C134. Patients will also be followed with MRI scans for potential clinical response to C134. The clinical strategy takes advantage of the virus' ability to infect and kill tumor cells while making new virus within the tumors cells; a critical enhancement of this effect is accomplished by the induction of an anti-tumor immune response; both effects are produced by the IRS-1 gene that was placed into the virus by genetic engineering. An additional important component of the research are systematic assessments of the quality of life on treated patients.

DETAILED DESCRIPTION:
The efficacy of herpes simplex virus (HSV) as a treatment for brain tumors has been demonstrated experimentally. The earliest studies used an HSV that was genetically engineered so that the gene for an important enzyme, thymidine kinase (tk) was deleted. This engineered virus still killed tumor cells but was not toxic. Martuza and colleagues demonstrated that tumors implanted in mice shrank following treatment with varying doses of this virus.

Additional modified viruses based on the HSV backbone have been developed and tested with encouraging results.Viruses containing deletions in other important viral genes (e.g., DNA polymerase and the gene which can make the virus neurotoxic, γ134.5), also retained the capability of killing cultured human tumors but did not injure mice; in particular, they were safe for use in the brain. These viruses retained the viral tk gene, and so are susceptible to the antiviral drug acyclovir which is routinely used to treat HSV Infection, making them even more safe .

Martuza and colleagues generated G207, a modified HSV that contains (1) deletions of both copies of γ134.5 and (2) another gene called ribonucleotide reductase, was disabled secondary to disruption of the U139 gene by insertion of the E. coli LacZ coding region . G207 significantly prolonged survival of nude mice bearing human tumors. In addition, virus injected into the brains of the HSV sensitive primates (Aotus) did not produce any deleterious side effects.

G207 and 1716 have both been used in human trials. A dose-escalating phase 1 study of G207 was completed in patients with recurrent, progressive malignant glioma . The trial was conducted at University of Alabama at Birmingham and Georgetown University Medical Center. Twenty-one patients were enrolled in a total of seven dose-escalating cohorts, with three patients per cohort. Patients were stereotactically inoculated with G207 in the enhancing portions of their tumors. Five separate loci were inoculated in the final cohort; all previous cohorts were inoculated in a single locus within the enhancing tissue only. No toxicity definitively related to G207 was observed at doses up to 3 x 109 plaque forming units (pfu-these are active viral particles). In fact, a toxic dose level was not attained during this trial. This was due to viral processing techniques, limiting the total dose that could be administered.

In a Phase IB study, six patients with recurrent, resectable malignant glioma were enrolled at the University of Alabama at Birmingham, in a trial examining a split dose administration strategy of G207. Patients underwent inoculation of G207 into their tumors, followed two to five days later by resection of the tumor and reinoculation of G207 into the tumor cavity. No dose limiting toxicities were seen in the trial, although one patient suffered a twelve hour period of mental status changes, weakness, and an elevated temperature when a protocol deviation resulted in an inadvertent partial dose of virus being administered intraventricularly, into the cerebrospinal fluid chamber of the brain. The patient fully recovered quickly and fully. One of the six patients went nearly two years before remote recurrence of her glioblastoma multiforme resulted in her death. A third study in 9 patients with recurrent malignant glioma was completed in which G207 was being administered followed by a single small dose of 5Gy of radiation. Nine patients were followed without any dose limiting toxicity, and some patients had remarkable responses to treatment. Currently, two clinical studies of oncolytic HSV are underway that examine G207 in pediatric patients as well as a novel oncolytic HSV expressing IL- 12, in adult patients. No findings of these two studies have yet been reported.

C134 was designed to replicate better than 1st gen HSVs. C134 is created by by inserting the PKR evasion gene, IRS1. from an evolutionary distant herpesvirus HCMV, which allows the virus to replicate much better but does not produce toxicity.

The described G207 trials clearly demonstrate that increased immune cell infiltrates within MG are associated with better outcomes. C134 elicits a robust immune response that contributes greatly to its antitumor effects.

C134 combines advantages of both wild-type and Δγ134.5 HSV and is an improvement over 1st generation viruses. C134 replicates and lyses tumor cells like a wild-type HSV in the IFN aberrant tumor environment, but is safe in normal cells. C134 induces immune responses which exceed those produced by 1st generation viruses. The study is designed to use all the information from any patients already treated to determine what the best dose for the next patient should be.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed recurrent/progressive glioblastoma multiforme, anaplastic astrocytoma, or gliosarcoma.
* Prior therapy. Patients must have failed external beam radiotherapy to the brain at least 4 weeks prior to enrollment.
* Age 18 years or older, because no dosing or adverse event data are currently available on the use of IRSl-chimeric HSVl in patients below 18 years of age, children are excluded from this study but will be eligible for future pediatric phase 1 single-agent trials. Note: 18 is the age of majority in the state of Alabama for participation in clinical trials.
* Karnofsky Performance Status ≥70%
* Life expectancy of greater than 4 weeks.
* Patients must have normal organ and marrow function as defined below:

  * leukocytes ≥3,000/uL
  * absolute neutrophil count ≥1,500/uL
  * platelets ≥100,000/uL
  * total bilirubin within normal institutional limits
  * AST(SGOT)/ ALT(SGPT) ≤2.5 X institutional upper limit of normal
  * Creatinine within normal institutional limits OR Creatinine clearance ≥60 mL/min/1.73 m2 for patients with creatinine levels
* Residual lesion must be ≥1.0 and < 5.5 cm in diameter without bilateral extension through the corpus callosum as determined by MRI as this is a locally delivered treatment. These parameters will be re-evaluated on imaging done on the day of catheter implantation and if the lesion no longer meets the criteria, the patient will not undergo catheter implantation or treatment with C134.
* The effects of IRS1-chimeric HSV1 on the developing human fetus are unknown. For this reason, women of child-bearing potential and men must agree to use adequate contraception prior to study entry and for the first six months after receiving IRS1-chimeric HSVl. Because it is currently unknown if IRS1-chimeric HSV1 can be transmitted by sexual contact, a barrier method of birth control should be employed. Should a woman become pregnant while participating in this study, she should inform her treating physician immediately.
* Ability to understand and the willingness to sign a written informed consent document (Informed consent document in Appendix E).
* Females of childbearing potential must not be pregnant; this will be confirmed by a negative serum pregnancy test within 14 days prior to starting study treatment.
* Steroid use is allowed as long as dose has not increased within 2 weeks of scheduled C134 administration whenever possible, the patient should be on a steroid dose that is equivalent to a dexamethasone dose of ≤2mg daily at the time of treatment.

Exclusion Criteria:

* Patients who have had chemotherapy, cytotoxic therapy, immunotherapy or gene therapy within 6 weeks prior to entering the study, surgical resection within 4 weeks prior to entering the study, or have received experimental viral therapy at any time (e.g., adenovirus, retrovirus or herpesvirus * protocol). Also, those who have not recovered from adverse events due to therapeutic interventions administered more than 4 weeks earlier.
* Patients may not be receiving any other investigational agents.
* History of allergic reactions attributed to compound of similar biologic composition to IRS1-chimeric HSVl.
* Tumor involvement which would require ventricular, brainstem, basal ganglia, or posterior fossa inoculation or would require access through a ventricle in order to deliver treatment.
* Prior history of encephalitis, multiple sclerosis, or other CNS infection.
* Required steroid increase within 2 weeks of scheduled IRS1-chimeric HSV1 administration.
* Active oral herpes lesion.
* Concurrent therapy with any drug active against HSV (acyclovir, valaciclovir, penciclovir, famciclovir, ganciclovir, foscarnet, cidofovir).
* Uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or any other medical condition that precludes surgery . Also, psychiatric illness/social situations that would limit compliance with study requirements.
* Required steroid increase within 2 weeks of scheduled C134 administration. When possible, the patient should be on a dexamethasone equivalent dose of ≤2mg daily at the time of treatment.
* Known history of allergic reaction to IV contrast material that is not amenable to pre-treatment by UAB protocol.
* Have a pacemaker, ferro-magnetic aneurysm clips, metal infusion pumps, metal or shrapnel fragments, or certain types of stents.
* Received Bevacizumab (Avastin) therapy within 4 weeks of scheduled C134 administration.
* Excluded patient groups

  * Pregnant women are excluded from this study because IRS1-chimeric HSV1 is a viral oncolytic therapy with unknown potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with IRS1-chimeric HSV1, breastfeeding should be discontinued if the mother is treated with IRS1-chimeric HSVl.
  * Because patients with immune deficiency will be unable to mount the anticipated immune response underlying this therapeutic rationale, HIV-seropositive patients are excluded from this study. Other treatment studies for this disease that are less dependent on the patients' immune response are more appropriate for HIV-seropositive patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2019-09-23 (Actual); Primary Completion 2024-10-25 (Actual); Study Completion 2026-09 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: James Markert, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- 10^6 Single Dose of C134: Participants were administered 10^6 single dose of C134 infused through catheters into region(s) of tumor defined by MRI
- 10^7 Single Dose of C134: Participants were administered 10^7 single dose of C134 infused through catheters into region(s) of tumor defined by MRI
- 10^7.5 Single Dose of C134: Participants were administered 10^7.5 single dose of C134 infused through catheters into region(s) of tumor defined by MRI
- 10^5 Single Dose of C134: Participants were administered 10^5 single dose of C134 infused through catheters into region(s) of tumor defined by MRI
- 10^5.5 Single Dose of C134: Participants were administered 10^5.5 single dose of C134 infused through catheters into region(s) of tumor defined by MRI
- Screen Fails: Participants that consented to the study, but ended up becoming ineligible before they were given C134
Period: Overall Study
Arm/Group | 10^6 Single Dose of C134 | 10^7 Single Dose of C134 | 10^7.5 Single Dose of C134 | 10^5 Single Dose of C134 | 10^5.5 Single Dose of C134 | Screen Fails
Started | 2 | 2 | 1 | 8 | 1 | 5
Completed | 1 | 0 | 0 | 1 | 1 | 0
Not Completed | 1 | 2 | 1 | 7 | 0 | 5
Not completed — Death | 0 | 1 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Screen Fail | 0 | 0 | 0 | 0 | 0 | 5
Not completed — Disease Progression | 1 | 1 | 0 | 5 | 0 | 0
Not completed — Insurance Coverage | 0 | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 10^6 Single Dose of C134 | 10^7 Single Dose of C134 | 10^7.5 Single Dose of C134 | 10^5 Single Dose of C134 | 10^5.5 Single Dose of C134 | Screen Fails | Total
Number analyzed (Participants) | 2 | 2 | 1 | 8 | 1 | 5 | 19
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 2 | 1 | 1 | 6 | 1 | 4 | 15
  >=65 years | 0 | 1 | 0 | 2 | 0 | 1 | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 0 | 3 | 1 | 3 | 8
  Male | 1 | 2 | 1 | 5 | 0 | 2 | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 2 | 2 | 1 | 8 | 1 | 5 | 19
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: Participants]
  United States | 2 | 2 | 1 | 8 | 1 | 5 | 19

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose of C134 Treatment
Description: Dose modifications will utilize a modified Continual Reassessment Method (CRM) for each successive subject until an MTD or the maximal planned dose is reached.
Time Frame: from baseline through month 12
Measure: Number; unit: Plaque-forming units (PFU)
Arm/Group | C134 Treatment
Number analyzed (Participants) | 14
Plaque-forming units (PFU) | 31,622,776.6

2. Secondary Outcome: Measure of Progression Free Survival
Description: Patients will receive contrast-enhanced MRI to monitor progression (changes in tumor volume or tumor enhancement assessed by the iRANO criteria). As indicated in the criteria, biopsy and/or resection may be performed in instances of uncertainty. Determination of time to progression (in months) will be recorded for each patient and median progression-free survival will be calculated for the entire cohort (Kaplan-Meier).
Time Frame: pre-study, day 3, day 28, month 3, month 6, month 12
Reporting Status: Not Posted

3. Secondary Outcome: Measure Overall Survival
Description: Patients survival will be recorded (Kaplan-Meier).
Time Frame: day 0, day 1, day 2, day 3, day 7, day 28, month 3, month 6, month 12
Reporting Status: Not Posted

4. Secondary Outcome: Measurement of HSV Titer
Description: Detection and quantification of HSV antibody titer via ELISA, pfu/mL.
Time Frame: pre-study, day 28, month 3, month 6, month 12
Reporting Status: Not Posted

5. Secondary Outcome: Composition of the White Blood Cells
Description: White blood cell subset analysis by FACS, as a percent of total white blood cell number.
Time Frame: pre-study, day 2, day 7, day 28, month 3, month 6, month 12
Reporting Status: Not Posted

6. Secondary Outcome: Measure Interferon Levels
Description: Intracellular lymphocyte interferon levels will be assessed by FACS analysis ng/mL
Time Frame: pre-study, day 2, day 7, day 28, month 3, month 6, month 12
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 12 Months
Description: Adverse events were not collected for participants listed under "Screen Fails". Participants in this group were enrolled, but withdrawn from the study for various reasons, prior to administration of the the study drug.
Arm/Group | 10^6 Single Dose of C134 | 10^7 Single Dose of C134 | 10^7.5 Single Dose of C134 | 10^5 Single Dose of C134 | 10^5.5 Single Dose of C134
All-Cause Mortality (participants affected / at risk) | 2/2 | 2/2 | 1/1 | 6/8 | 0/1
Serious Adverse Events (participants affected / at risk) | 2/2 | 2/2 | 1/1 | 7/8 | 1/1
Other Adverse Events (participants affected / at risk) | 2/2 | 2/2 | 1/1 | 8/8 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 10^6 Single Dose of C134 (N=2) | 10^7 Single Dose of C134 (N=2) | 10^7.5 Single Dose of C134 (N=1) | 10^5 Single Dose of C134 (N=8) | 10^5.5 Single Dose of C134 (N=1)
Neurological (Nervous system disorders) | 2 (3) | 1 (3) | 1 (3) | 7 (11) | 1 (3)
Respiratory (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sensory (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Cardiovascular (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
HEENT (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hematology/Lymphatic (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 10^6 Single Dose of C134 (N=2) | 10^7 Single Dose of C134 (N=2) | 10^7.5 Single Dose of C134 (N=1) | 10^5 Single Dose of C134 (N=8) | 10^5.5 Single Dose of C134 (N=1)
Acalculia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute mastoiditis of right side (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
A-Fib (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Aphasia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Appetite, dry heaves (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aspiration Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ataxia of left arm (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cataracts bilateral (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cerebral edema (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Collapsed at work, did not lose consciousness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Confused and difficulty with productive speech CTH (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CSF positive candida (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
CSF positive for HSV (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Decreased cognitive processing (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Decreased mobility-barely able to walk from room to room with assistance (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Decreased visual acuity (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Depressed mood (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Difficulty sleeping (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diplopia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Disease progression (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dry skin, patches (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ear pain, right side (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Elevated Blood Pressure (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Elevated temperature (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Encephilitis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Eye disorders (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Fall (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Febrile (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Feels "Loopy" (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fever (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
GBM growth /Increased tumor size (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
General deconditioning (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 5 (6) | 0 (0)
Hearing decreased (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hemotoma (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperglycemia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypersensitivity to smell (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Increased agitation (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Increased intracranial pressure (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Increased sleepiness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Increased somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Increased tremors of extremities (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Increased weakness Right side (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intermittent confusion (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Left homonymous VF defect (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Left sided weakness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lethargy/energy crash (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Loss of appetite (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Low grade temperature (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Memory impairment (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mild cognitive symptoms (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Mild syncope when standing from sitting (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Morbilliform drug eruption rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Slight increase in enhancing, moderate increase vasogenic edema (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Increased enhancement, edema and mass effect (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Multiple blood clots in chest in legs (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Muscle weakness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (3) | 0 (0)
Nodule of enhancement concerning for tumor progression (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Not able to communicate, either words not understandable or won't answer questions (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Numbness in right foot and lower leg (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oral PCR positive for HSV (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Overall decline in subject's status, Hospice initiated (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain in right tonsil (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Personality change (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Photophobia (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Progression of malignant neoplasm (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Partial seizures (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pulmonary embolus (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Repetitive activities (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Retinopathy (bilateral retinitis) (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash on face (after shaving) (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Right facial muscle weakness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Seizures (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Serum Calcium lab value decreased (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Serum draw on 9/20 reported Positive for HSV CPT (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Severe headache with nausea (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Short term memory loss (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Significant somatosensory dysfunction to left body (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin infection (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin lesions (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Slurred speech (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Small amount of pneumocephalus on CTH (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Somnolent (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Spasticity right sided, worse in upper extremity (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Stumble and fall X3 (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thrombus in cephalic veins bilaterally (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tumor progression (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Unresponsive/Obtunded - intubated (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinalysis with trace LE (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1)
Vision decreased (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Visual disturbances (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vitreous detachment (floaters) (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Weakness and dystonia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Worsened dysphasia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Worsening ataxia (foot drag) (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Worsening cognitive symptoms (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Worsening speech (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Hypernatremia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2023-12-17): https://cdn.clinicaltrials.gov/large-docs/76/NCT03657576/Prot_SAP_ICF_000.pdf